CLINICAL TRIAL: NCT04069481
Title: Dance for the Improvement of Balance and Gait After Stroke: A Randomized Controlled Trial
Brief Title: Dance for the Improvement of Balance and Gait After Stroke
Acronym: DASRCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Kara Patterson, Scientist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G-17-0018263
Record Dates: First submitted 2019-08-07; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Chronic Stroke
Keywords: Dance; Stroke; Randomized Controlled Trial; Rehabilitation; Gait; Balance
MeSH Terms: conditions — Stroke | interventions — Mindfulness; Exercise; Control Groups

STUDY DESIGN:
Intervention Model Description: Two groups of participants. One group receives the dance intervention. The control group will receive mindful meditation, strengthening & stretching exercises.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dance intervention (Experimental): Participants will receive a 1-hour group dance class twice a week for 12 weeks. Classes will include a seated warm up, dance exercises in standing, dance activities moving across the floor, throughout the space and conclude with a bow exercise. Music and dance styles will vary and personal preference of participants will also be taken into account.
  Interventions: Other: Dance
- Exercise and mindfulness meditation (Active Comparator): Participants will receive a 1-hour group exercise class twice a week for 12 weeks. Classes will include resistance training exercises with resistance bands, stretching and range of motion exercises in seated and standing positions. Classes will also include mindfulness exercises. During active exercises music will be played and personal preference of participant will be taken into account.
  Interventions: Other: Mindfulness meditation and Exercise

INTERVENTIONS:
Other: Dance — One-hour class, twice a week. Classes include dance warm up exercises, various dance movements and choreography that include coordinated whole body movements through space synchronized to music.
  Other Names: Intervention group
  Arms: Dance intervention
Other: Mindfulness meditation and Exercise — One hour class, twice a week. Classes include upper and lower extremity stretching and resistance exercises and mindfulness meditation, that includes body scan technique and breathing exercises.
  Other Names: Control group
  Arms: Exercise and mindfulness meditation

SUMMARY:
Stroke can drastically impact the ability to walk and keep your balance. In addition people with chronic stroke feel social isolated, become less satisfied with their walking and lose confidence in their ability to move without falling.

Ned new treatments are needed for walking and balance. Dancing is a fun, social activity that has similar benefits to traditional exercise. Another benefit of dancing is the use of music, which improves mood, increases motivation and can even improve motor performance. Finally, moving in synchrony with other people during dancing can make people feel connected. We believe that dance classes can benefit people with stroke, but few studies have been done.

The objective of our project is to conduct a randomized controlled trial to test whether dance can improve balance and walking for people with chronic stroke. The investigators are also interested in whether dancing improves people's confidence in their ability to do activities without losing their balance (i.e. balance confidence), decreases their feelings of isolation and increases their quality of life.

DETAILED DESCRIPTION:
This study is a randomized controlled trial to investigate the effects of an adapted dance program for people with chronic stroke. Participants with stroke living in the community will be randomly assigned to either the dance group or the control group. Participants will attend classes 2 times a week for 12 weeks. The primary outcomes are change in balance balance (measured with the Mini BESTest) and change in gait speed. Participants will be assessed before and after the 12 week program.

ELIGIBILITY:
Inclusion Criteria:

1. > 6 months post stroke
2. Ability to transfer sit to stand and stand to sit with minimal use of arm rests
3. Ability to stand without physical support from an aid or another person for 30 seconds
4. Ability to walk 10m without physical assistance from a walking device, but with standby assistance from another person if needed
5. Ability to follow 2-3 step instructions with minimal prompting from another person
6. Have received clearance from their physician to participate in exercise.

Exclusion Criteria:

1. Severe hearing loss
2. Pre-existing conditions that significantly impact gait and balance (e.g. osteoarthritis)
3. Other neurological conditions that impact gait and balance (e.g. PD).
4. Have participated in a dance class within the past 12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in balance | at study completion on average 14 weeks
  Mini-Balance Evaluation Systems Test (Mini-BESTest)
  The Mini-BESTest is a 14-item performance-based clinical scale that will be used to measure balance during standing and walking activities. There are 4 subscales in the miniBESTest and the scores on the subscales are summed to create the total score. The miniBESTest total score can range form 0-56 and higher scores indicate better balance. The Mini-BESTest shows good inter- (ICC 0.96) and intra-rater (ICC=0.97) and test-retest reliability (ICC=0.98) in the stroke population.
Change in gait speed | at study completion on average 14 weeks
  Gait speed will be measured in m/sec with a with a pressure sensitive mat

SECONDARY OUTCOMES:
Change in social isolation | at study completion on average 14 weeks
  Friendship scale
  The Friendship scale is a short (6-item) and user-friendly measure of perceived social isolation developed for older adults. It has a maximum score of 24 and lower scores indicate higher levels of social isolation. It has internal structure (RMSEA=0.02) and reliability (Chronbach α=0.83)
Change in Quality of life scale | at study completion on average 14 weeks
  Stroke Specific Quality Of Life scale (SS-QOL)
  The SS-QOL is a self-report scale containing 49 items in 12 domains ranging from mobility and energy to mood and language. The SS-QOL has both domain scores and an overall SS-QOL summary score. The domain scores are unweighted averages of the associated items while the summary score is an unweighted average of all twelve domain scores. The scores can range from 0 to 5 and higher scores indicate better quality of life.
  The SS-QOL had good internal consistency (range Chronbach α=0.75-0.89), test-retest reliability (r=0.92) and inter-rater reliability (r=0.92).
Change in balance confidence | at study completion on average 14 weeks
  Activity Balance Confidence Scale (ABC)
  The ABC is a 16-item self-report scale that requires individuals indicate their confidence in performing various activities without losing their balance or becoming unsteady. The ABC total score is calculated as an average of the ratings for the 16 items. The score ranges from 0-100 and higher scores indicate greater confidence. The ABC scale has good internal consistency (α=0.94) and test-retest reliability (ICC =0.85) in individuals with chronic stroke living in the community
Change in upper extremity active range of motion (AROM) | at study completion on average 14 weeks
  active range of motion of the shoulder assessed using a measuring tape and a ruler to quantify arm elevation, lateral rotation and medial rotation.

CONTACTS AND LOCATIONS:
Overall Officials: Kara Patterson, PhD, Principal Investigator — Toronto Rehabilitation/ University of Toronto; Dina Brooks, PhD, Principal Investigator — Toronto Rehabilitation
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available.

REFERENCES:
- [Background] Tsang CS, Liao LR, Chung RC, Pang MY. Psychometric properties of the Mini-Balance Evaluation Systems Test (Mini-BESTest) in community-dwelling individuals with chronic stroke. Phys Ther. 2013 Aug;93(8):1102-15. doi: 10.2522/ptj.20120454. Epub 2013 Apr 4. PMID 23559522
- [Background] Wong JS, Jasani H, Poon V, Inness EL, McIlroy WE, Mansfield A. Inter- and intra-rater reliability of the GAITRite system among individuals with sub-acute stroke. Gait Posture. 2014;40(1):259-61. doi: 10.1016/j.gaitpost.2014.02.007. Epub 2014 Feb 26. PMID 24630463
- [Background] Patterson KK, Gage WH, Brooks D, Black SE, McIlroy WE. Changes in gait symmetry and velocity after stroke: a cross-sectional study from weeks to years after stroke. Neurorehabil Neural Repair. 2010 Nov-Dec;24(9):783-90. doi: 10.1177/1545968310372091. Epub 2010 Sep 14. PMID 20841442
- [Background] Garland SJ, Willems DA, Ivanova TD, Miller KJ. Recovery of standing balance and functional mobility after stroke. Arch Phys Med Rehabil. 2003 Dec;84(12):1753-9. doi: 10.1016/j.apmr.2003.03.002. PMID 14669179
- [Background] Hawthorne G Measuring social isolation in older adults: development and initial validation of the friendship scale. Social Indicators Research 2006; 77: 521-548
- [Background] Williams LS, Weinberger M, Harris LE, Clark DO, Biller J. Development of a stroke-specific quality of life scale. Stroke. 1999 Jul;30(7):1362-9. doi: 10.1161/01.str.30.7.1362. PMID 10390308
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Botner EM, Miller WC, Eng JJ. Measurement properties of the Activities-specific Balance Confidence Scale among individuals with stroke. Disabil Rehabil. 2005 Feb 18;27(4):156-63. doi: 10.1080/09638280400008982. PMID 15824045
- [Background] Uswatte G, Taub E, Morris D, Vignolo M, McCulloch K. Reliability and validity of the upper-extremity Motor Activity Log-14 for measuring real-world arm use. Stroke. 2005 Nov;36(11):2493-6. doi: 10.1161/01.STR.0000185928.90848.2e. Epub 2005 Oct 13. PMID 16224078
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Patterson KK, Wong JS, Nguyen TU, Brooks D. A dance program to improve gait and balance in individuals with chronic stroke: a feasibility study. Top Stroke Rehabil. 2018 Sep;25(6):410-416. doi: 10.1080/10749357.2018.1469714. Epub 2018 May 10. PMID 29745307